CLINICAL TRIAL: NCT01928771
Title: A Multicentre, Randomized, Double-blind, Parallel Group, Placebo-controlled, Phase III Efficacy and Safety Study of Benralizumab (MEDI-563) Added to High-dose Inhaled Corticosteroid Plus Long-acting β2 Agonist in Patients With Uncontrolled Asthma
Brief Title: Efficacy and Safety Study of Benralizumab Added to High-dose Inhaled Corticosteroid Plus LABA in Patients With Uncontrolled Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3250C00017
Record Dates: First submitted 2013-08-16; First posted 2013-08-27 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Asthma,; Bronchial Diseases,; Respiratory Tract Diseases,; Lung Diseases,; Obstructive Lung Diseases
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Benralizumab 30 mg q.4 weeks (Experimental): Benralizumab administered subcutaneously every 4 weeks
  Interventions: Biological: Benralizumab
- Benralizumab 30 mg q.8 weeks (Experimental): Benralizumab administered subcutaneously every 8 weeks
  Interventions: Biological: Benralizumab
- Placebo (Placebo Comparator): Placebo administered subcutaneously
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Benralizumab — Benralizumab subcutaneously on study week 0 until study week 44 inclusive.
  Arms: Benralizumab 30 mg q.4 weeks; Benralizumab 30 mg q.8 weeks
Biological: Placebo — Placebo subcutaneously on study week 0 until study week 44 inclusive.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Benralizumab reduces the number of asthma exacerbations in patients who remain uncontrolled on high doses of ICS-LABA.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for study participation must be obtained prior to any study related procedures being performed (local regulations are to be followed in determining the assent/consent requirements for children and parent[s]/guardian[s]) and according to international guidelines and/or applicable European Union guidelines.
2. Female and Male aged 12 to 75 years inclusively, at the time of visit 1. For those patients, who are 17 on the day of Visit 1 but will turn 18 after this day, will be considered an adolescent for the purposes of this trial.
3. History of physician-diagnosed asthma requiring treatment with medium-to-high dose ICS (>250μg fluticasone dry powder formulation equivalents total daily dose) and a LABA, for at least 12 months prior to Visit 1
4. Documented treatment with ICS and LABA for at least 3 months prior to Visit 1 with or without oral corticosteroids and additional asthma controllers.

   * For subjects 18 years of age and older, the ICS dose must be >500 mcg/day fluticasone propionate dry powder formulation or equivalent daily.
   * For subjects ages 12-17, the ICS dose must be ≥500 mcg /day fluticasone propionate dry powder formulation or equivalent daily.

Exclusion criteria:

1. Clinically important pulmonary disease other than asthma (e.g. active lung infection, COPD, bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha 1 anti-trypsin deficiency, and primary ciliary dyskinesia) or ever been diagnosed with pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil counts (e.g. allergic bronchopulmonary aspergillosis/mycosis, Churg- Strauss syndrome, hypereosinophilic syndrome)
2. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could:

   * Affect the safety of the patient throughout the study
   * Influence the findings of the studies or their interpretations
   * Impede the patient's ability to complete the entire duration of study
3. Acute upper or lower respiratory infections requiring antibiotics or antiviral medication within 30 days prior to the date informed consent is obtained or during the screening/run-in period
4. Any clinically significant abnormal findings in physical examination, vital signs, haematology, clinical chemistry, or urinalysis during screening/run-in period, which in the opinion of the Investigator, may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or the patient's ability to complete entire duration of the study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2681 (Actual)
Dates: Start 2013-09-19; Primary Completion 2016-04-05 (Actual); Study Completion 2016-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene R. Bleecker, MD, Professor of Medicine, Principal Investigator — Center for Genomics and Personalized Medicine Research, Medical Center Boulevard, Winston-Salem, North Carolina 27157
Locations (275):
- United States (110):
  - Research Site, Foley, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Scottsboro, Alabama
  - Research Site, Sheffield, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Beverly Hills, California
  - Research Site, Costa Mesa, California
  - Research Site, Huntington Beach, California
  - Research Site, Huntington Park, California
  - Research Site, Los Angles, California
  - Research Site, Newport Beach, California
  - Research Site, Orange, California
  - Research Site, Riverside, California
  - Research Site, San Jose, California
  - Research Site, Santa Ana, California
  - Research Site, Hartford, Connecticut
  - Research Site, New Haven, Connecticut
  - Research Site, Brandon, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Cutler Bay, Florida
  - Research Site, DeLand, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Homestead, Florida
  - Research Site, Jackonsville, Florida
  - Research Site, Lynn Haven, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Sebring, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Albany, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Gurnee, Illinois
  - Research Site, Normal, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Fort Mitchell, Kentucky
  - Research Site, Hazard, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Opelousas, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Gardner, Massachusetts
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Quincy, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Picayune, Mississippi
  - Research Site, Billings, Montana
  - Research Site, Bellevue, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Sparks, Nevada
  - Research Site, Marlton, New Jersey
  - Research Site, Northfield, New Jersey
  - Research Site, Union, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Hopewell Jct, New York
  - Research Site, New York, New York
  - Research Site, Staten Island, New York
  - Research Site, The Bronx, New York
  - Research Site, Huntersville, North Carolina
  - Research Site, Shelby, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Grand Forks, North Dakota
  - Research Site, Oregon, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Wooster, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Erie, Pennsylvania
  - Research Site, Feasterville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Phoenixville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Warwick, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Easley, South Carolina
  - Research Site, Hodges, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Germantown, Tennessee
  - Research Site, Allen, Texas
  - Research Site, Dallas, Texas
  - Research Site, Dickinson, Texas
  - Research Site, Duncanville, Texas
  - Research Site, Georgetown, Texas
  - Research Site, Houston, Texas
  - Research Site, McAllen, Texas
  - Research Site, McKinney, Texas
  - Research Site, Pharr, Texas
  - Research Site, Plano, Texas
  - Research Site, Sealy, Texas
  - Research Site, Splendora, Texas
  - Research Site, Orem, Utah
  - Research Site, Provo, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Abingdon, Virginia
  - Research Site, Hopewell, Virginia
  - Research Site, Morgantown, West Virginia
  - Research Site, Greenfield, Wisconsin
- Australia (11):
  - Research Site, Bedford Park
  - Research Site, Box Hill
  - Research Site, Clayton
  - Research Site, Concord
  - Research Site, Frankston
  - Research Site, Nedlands
  - Research Site, New Lambton Heights
  - Research Site, Parkville
  - Research Site, Prahran
  - Research Site, Randwick
  - Research Site, Woolloongabba
- Brazil (5):
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santo André
  - Research Site, São Paulo
  - Research Site, Sorocaba
- Bulgaria (11):
  - Research Site, Dupnitsa
  - Research Site, Pernik
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Samokov
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Velingrad
  - Research Site, Yambol
- Czechia (10):
  - Research Site, Brno
  - Research Site, Jindřichův Hradec
  - Research Site, Karlovy Vary
  - Research Site, Ostrava
  - Research Site, Pardubice
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Rokycany
  - Research Site, Strakonice
  - Research Site, Teplice
- France (14):
  - Research Site, Brest
  - Research Site, Clermont-Ferrand
  - Research Site, Dijon
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Le Mans
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Pringy
  - Research Site, Saint-Pierre
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Italy (17):
  - Research Site, Bari
  - Research Site, Bologna
  - Research Site, Catania
  - Research Site, Cona
  - Research Site, Florence
  - Research Site, Foggia
  - Research Site, Legnago
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, San Pietro Vernotico
  - Research Site, Torino
  - Research Site, Verona
- Mexico (3):
  - Research Site, Guadalajara
  - Research Site, Monterrey
  - Research Site, Morelia
- Peru (3):
  - Research Site, Cusco
  - Research Site, Lima
  - Research Site, Surco
- Poland (16):
  - Research Site, Bialystok
  - Research Site, Dobre Miasto
  - Research Site, Gdansk
  - Research Site, Giżycko
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Kościan
  - Research Site, Legnica
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Proszowice
  - Research Site, Rzeszów
  - Research Site, Sosnowiec
  - Research Site, Wołomin
  - Research Site, Wroclaw
  - Research Site, Zgierz
- Russia (20):
  - Research Site, Chelyabinsk
  - Research Site, Ivanovo
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Pyatigorsk
  - Research Site, Rostov-on-Don
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Smolensk
  - Research Site, StPetersburg
  - Research Site, Tomsk
  - Research Site, Vladikavkaz
  - Research Site, Vladimir
  - Research Site, Volgograd
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- South Africa (5):
  - Research Site, Benoni
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, KwaDukuza
  - Research Site, Mowbray
- South Korea (9):
  - Research Site, Anyang-si
  - Research Site, Bucheon-si
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Jeju City
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (9):
  - Research Site, Barcelona
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Palma de Mallorca
  - Research Site, Sagunto(Valencia)
  - Research Site, Salamanca
  - Research Site, Valencia
- Turkey (Türkiye) (8):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Bursa
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kocaeli
  - Research Site, Mersin
- United Kingdom (22):
  - Research Site, Birmingham
  - Research Site, Bradford
  - Research Site, Cambridge
  - Research Site, Chertsey
  - Research Site, Chester
  - Research Site, Chippenham
  - Research Site, Cottingham
  - Research Site, Darlington
  - Research Site, Glasgow
  - Research Site, High Heaton/Newcastle Upon Tyn
  - Research Site, Leeds
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Maidstone
  - Research Site, Manchester
  - Research Site, Nottingham
  - Research Site, Plymouth
  - Research Site, Portsmouth
  - Research Site, Soham
  - Research Site, Somerset
  - Research Site, Stevenage
  - Research Site, Stockton
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

REFERENCES:
- [Derived] Menzies-Gow A, Hoyte FL, Price DB, Cohen D, Barker P, Kreindler J, Jison M, Brooks CL, Papeleu P, Katial R. Clinical Remission in Severe Asthma: A Pooled Post Hoc Analysis of the Patient Journey with Benralizumab. Adv Ther. 2022 May;39(5):2065-2084. doi: 10.1007/s12325-022-02098-1. Epub 2022 Mar 14. PMID 35287231
- [Derived] Lugogo NL, Kreindler JL, Martin UJ, Cook B, Hirsch I, Trudo FJ. Blood eosinophil count group shifts and kinetics in severe eosinophilic asthma. Ann Allergy Asthma Immunol. 2020 Aug;125(2):171-176. doi: 10.1016/j.anai.2020.04.011. Epub 2020 Apr 22. PMID 32334141
- [Derived] Jackson DJ, Humbert M, Hirsch I, Newbold P, Garcia Gil E. Ability of Serum IgE Concentration to Predict Exacerbation Risk and Benralizumab Efficacy for Patients with Severe Eosinophilic Asthma. Adv Ther. 2020 Feb;37(2):718-729. doi: 10.1007/s12325-019-01191-2. Epub 2019 Dec 14. PMID 31836949
- [Derived] Chipps BE, Hirsch I, Trudo F, Alacqua M, Zangrilli JG. Benralizumab efficacy for patients with fixed airflow obstruction and severe, uncontrolled eosinophilic asthma. Ann Allergy Asthma Immunol. 2020 Jan;124(1):79-86. doi: 10.1016/j.anai.2019.10.006. Epub 2019 Oct 15. PMID 31626906
- [Derived] Chupp G, Lugogo NL, Kline JN, Ferguson GT, Hirsch I, Goldman M, Zangrilli JG, Trudo F. Rapid onset of effect of benralizumab on morning peak expiratory flow in severe, uncontrolled asthma. Ann Allergy Asthma Immunol. 2019 May;122(5):478-485. doi: 10.1016/j.anai.2019.02.016. Epub 2019 Feb 23. PMID 30802500
- [Derived] Bleecker ER, Wechsler ME, FitzGerald JM, Menzies-Gow A, Wu Y, Hirsch I, Goldman M, Newbold P, Zangrilli JG. Baseline patient factors impact on the clinical efficacy of benralizumab for severe asthma. Eur Respir J. 2018 Oct 18;52(4):1800936. doi: 10.1183/13993003.00936-2018. Print 2018 Oct. PMID 30139780
- [Derived] DuBuske L, Newbold P, Wu Y, Trudo F. Seasonal variability of exacerbations of severe, uncontrolled eosinophilic asthma and clinical benefits of benralizumab. Allergy Asthma Proc. 2018 Sep 4;39(5):345-349. doi: 10.2500/aap.2018.39.4162. Epub 2018 Aug 4. PMID 30077185
- [Derived] Chipps BE, Newbold P, Hirsch I, Trudo F, Goldman M. Benralizumab efficacy by atopy status and serum immunoglobulin E for patients with severe, uncontrolled asthma. Ann Allergy Asthma Immunol. 2018 May;120(5):504-511.e4. doi: 10.1016/j.anai.2018.01.030. Epub 2018 Feb 1. PMID 29409951
- [Derived] Bleecker ER, FitzGerald JM, Chanez P, Papi A, Weinstein SF, Barker P, Sproule S, Gilmartin G, Aurivillius M, Werkstrom V, Goldman M; SIROCCO study investigators. Efficacy and safety of benralizumab for patients with severe asthma uncontrolled with high-dosage inhaled corticosteroids and long-acting beta2-agonists (SIROCCO): a randomised, multicentre, placebo-controlled phase 3 trial. Lancet. 2016 Oct 29;388(10056):2115-2127. doi: 10.1016/S0140-6736(16)31324-1. Epub 2016 Sep 5. PMID 27609408
- See also: D3250C00017CSP3redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1845&filename=D3250C00017_Revised_CSP_SIROCCO.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2681 participants signed informed consent form, 2232 participants entered screening/run-in period,1205 participants were randomised to receive treatment with benralizumab 30 mg Q4W, Q8W, or placebo. Of the 1205 patients randomised, 1204 patients received treatment with the study drug.
Groups:
- Benralizumab 30 mg q.4 Weeks: Benralizumab administered every 4 weeks subcutaneously.
- Benralizumab 30 mg q.8 Weeks: Benralizumab administered every 8 weeks subcutaneously.
Period: Overall Study
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Started | 400 | 398 | 407
Received Treatment | 399 | 398 | 407
Completed | 354 | 358 | 367
Not Completed | 46 | 40 | 40
Not completed — Adverse Event | 6 | 5 | 1
Not completed — Death | 2 | 2 | 2
Not completed — Lost to Follow-up | 5 | 6 | 3
Not completed — Withdrawal by Subject | 20 | 15 | 17
Not completed — Study-Specific Withdrawal Criteria | 0 | 1 | 1
Not completed — Other Reasons | 9 | 9 | 14
Not completed — Severe Non-Compliance to Protocol | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo | Total
Number analyzed (Participants) | 399 | 398 | 407 | 1204
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.1 (13.4) | 47.6 (14.5) | 48.7 (14.9) | 48.8 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 252 | 269 | 796
  Male | 124 | 146 | 138 | 408

OUTCOME MEASURES:

1. Primary Outcome: Annual Asthma Exacerbation Rate in Adult and Adolescent Patients With Uncontrolled Asthma for Eosinophils >=300/uL
Description: The annual exacerbation rate is based on unadjudicated annual exacerbation rate reported by the investigator in the eCRF
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Least Squares Mean (95% Confidence Interval); unit: events/year
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 275 | 267 | 267
events/year | 0.73 [0.60 to 0.89] | 0.65 [0.53 to 0.80] | 1.33 [1.12 to 1.58]
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Negative binomial; Model includes covariates treatment group, region, number of exacerbations in the previous year, and use of maintenance oral corticosteroids; Rate ratio = 0.55, 95% CI 2-sided [0.42 to 0.71]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Negative binomial; [statistical method as in outcome 1, analysis 1]; Rate ratio = 0.49, 95% CI 2-sided [0.37 to 0.64]

2. Secondary Outcome: Annual Asthma Exacerbation Rate in Adult and Adolescent Patients With Uncontrolled Asthma for Eosinophils < 300/uL
Description: as for outcome 1
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils <300/uL
Measure: Least Squares Mean (95% Confidence Interval); unit: events/year
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 124 | 131 | 140
events/year | 0.85 [0.65 to 1.11] | 1.00 [0.78 to 1.28] | 1.21 [0.96 to 1.52]
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.047, Negative binomial; [statistical method as in outcome 1, analysis 1]; Rate ratio = 0.7, 95% CI 2-sided [0.5 to 1.0]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.268, Negative binomial; [statistical method as in outcome 1, analysis 1]; Rate ratio = 0.83, 95% CI 2-sided [0.59 to 1.16]

3. Secondary Outcome: Annual Asthma Exacerbation Rate Resulting Emergency Room Visits and Hospitalizations
Description: The annual exacerbation rate associated with an emergency room visit or a hospitalization (adjudicated)
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Least Squares Mean (95% Confidence Interval); unit: events/year
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 275 | 267 | 267
events/year | 0.11 [0.07 to 0.16] | 0.06 [0.04 to 0.11] | 0.18 [0.13 to 0.25]
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.053, Negative binomial; Model includes covariates treatment group, region, number of exacerbations resulting in ER/hospitalization in the previous year, and use of OCS; Rate ratio = 0.61, 95% CI 2-sided [0.37 to 1.01]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Negative binomial; [statistical method as in outcome 3, analysis 1]; Rate ratio = 0.37, 95% CI 2-sided [0.2 to 0.67]

4. Secondary Outcome: Number of Patients With >=1 Asthma Exacerbations
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Number; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 275 | 267 | 267
Participants | 100 (84.227) | 93 (72.002) | 135 (74.434)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Proportion of patients with >=1 asthma exacerbation; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for region, number of exacerbations in the previous year, use of OCS; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.37 to 0.78]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Proportion of patients with >=1 asthma exacerbation; Test type: Superiority or Other; p = 0.01, Cochran-Mantel-Haenszel; Controlling for region, number of exacerbations from the previous year, use of OCS; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.43 to 0.90]

5. Secondary Outcome: Time to First Asthma Exacerbation
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 275 | 267 | 267
Days | NA (84.227) [NA to NA] — Median time is not estimable due to less than 50% patients had exacerbations occurred. | NA (72.002) [NA to NA] — Median time is not estimable due to less than 50% patients had exacerbations occurred. | 300 (74.434) [199 to NA] — Upper 95% CI for median is not estimable due to the curve representing the upper confidence limit of the survival function is above 50%
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Time to first exacerbation; Test type: Superiority or Other; p < 0.001, Regression, Cox; Model includes treatment, number of exacerbations in the previous year, region, use of OCS; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.49 to 0.82]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Time to first exacerbation; Test type: Superiority or Other; p < 0.001, Regression, Cox; Model includes treatment, number of exacerbations from the previous year, region, use of OCS; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.46 to 0.78]

6. Secondary Outcome: Mean Change From Baseline to Week 48 in Pre-bronchodilator FEV1 (L) Value for Baseline Eosinophils >=300/uL
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinopiles >=300/uL
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 236 | 235 | 233
Liter | 0.353 (0.503) | 0.398 (0.546) | 0.237 (0.508)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis; Model includes treatment, baseline pre-BD FEV1, region, use of OCS, visit and treatment by visit; Mean Difference (Final Values) = 0.106, 95% CI 2-sided [0.016 to 0.196]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Model includes treatment, baseline pre-BD FEV1, region, use of OCS, visit and treatment by visit; Mean Difference (Final Values) = 0.159, 95% CI 2-sided [0.068 to 0.249]

7. Secondary Outcome: Mean Change From Baseline to Week 48 in Pre-bronchodilator FEV1 (L) Value for Baseline Eosinophils <300/uL
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinopiles <300/uL
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 105 | 119 | 125
Liter | 0.115 (0.417) | 0.238 (0.483) | 0.140 (0.4)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.644, Mixed Models Analysis; Model includes treatment, baseline pre-BD FEV1, region, use of OCS, visit and treatment by visit; Mean Difference (Final Values) = -0.025, 95% CI 2-sided [-0.134 to 0.083]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.057, Mixed Models Analysis; Model includes treatment, baseline pre-BD FEV1, region, use of OCS, visit and treatment by visit; Mean Difference (Final Values) = 0.102, 95% CI 2-sided [-0.003 to 0.208]

8. Secondary Outcome: Mean Change From Baseline to Week 48 in Asthma Symptom Score for Baseline Eosinophils >=300/uL
Description: Asthma symptoms during night time and daytime are recorded by the patient in the asthma daily diary. Symptom score values are from 0 (No asthma symptom) to 3 (unable to sleep because of asthma, or unable to do normal activities due to asthma), and total asthma symptom score is the sum of the daytime and night time score (0 to 6). Lower score (0) is indicating better asthma symptom, while higher score (6) is indicating worse asthma symptom. Baseline is defined as the average of data collected from the evening of study day -10 to the morning of study day 1. Each time point is calculated as bi-weekly means based on daily diary data. If more than 50% of scores are missing in a 14 day period then this is considered as missing. Symptom score lower is better.
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 197 | 178 | 180
Scores on a scale | -1.15 (1.31) | -1.34 (1.27) | -1.03 (1.07)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.442, Mixed Models Analysis; Model includes treatment, baseline asthma symptom score, region, use of OCS, visit and visit by treatment; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.27 to 0.12]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis; Model includes treatment, baseline asthma symptom score, region, use of OCS, visit and visit by treatment; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.45 to -0.06]

9. Secondary Outcome: Mean Change From Baseline to Week 48 in Asthma Symptom Score for Baseline Eosinophils <300/uL
Description: as for outcome 8
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils <300/uL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 93 | 91 | 99
Scores on a scale | -0.98 (1.19) | -1.04 (1.24) | -0.78 (0.99)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.169, Mixed Models Analysis; Model includes treatment, baseline asthma symptom score, region, use of OCS, visit and visit by treatment; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.48 to 0.08]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.043, Mixed Models Analysis; Model includes treatment, baseline asthma symptom score, region, use of OCS, visit and visit by treatment; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.57 to -0.01]

10. Secondary Outcome: Change in Asthma Rescue Medication
Description: Change from baseline to week 48 in number of rescue medication use (puffs/day)
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Mean (Standard Deviation); unit: Puffs/day
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 197 | 178 | 180
Puffs/day | -2.74 (4.29) | -2.78 (3.90) | -2.18 (4.38)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.1, Mixed Models Analysis; Model includes treatment, baseline asthma medication use, region, use of OCS, visit and visit by treatment; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-1.16 to 0.10]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.081, Mixed Models Analysis; Model includes treatment, baseline asthma medication use, region, use of OCS, visit and visit by treatment; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-1.21 to 0.07]

11. Secondary Outcome: Home Lung Function Assessment Based on Morning PEF
Description: Change from baseline to week 48 in home lung function morning peak expiratory flow [PEF]
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 205 | 181 | 189
L/min | 45.857 (84.227) | 36.994 (72.002) | 22.059 (74.434)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Morning PEF change from baseline to Week 48; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Model includes treatment, baseline morning PEF, region, use of OCS, visit and visit by treatment; Mean Difference (Final Values) = 23.32, 95% CI 2-sided [9.20 to 37.43]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Morning PEF change from baseline to Week 48; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis; Model includes treatment, baseline morning PEF, region, use of OCS, visit and visit by treatment; Mean Difference (Final Values) = 16.46, 95% CI 2-sided [2.08 to 30.83]

12. Secondary Outcome: Home Lung Function Assessment Based on Evening PEF
Description: Change from baseline to week 48 in home lung function evening peak expiratory flow [PEF]
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 203 | 187 | 189
L/min | 36.806 (86.271) | 33.460 (74.017) | 14.784 (68.799)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Evening PEF change from baseline to Week 48; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; Model includes treatment, baseline evening PEF, region, use of OCS, visit and visit by treatment; Mean Difference (Final Values) = 21.75, 95% CI 2-sided [7.86 to 35.65]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Evening PEF change from baseline to Week 48; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis; Model includes treatment, baseline evening PEF, region, use of OCS, visit and visit by treatment; Mean Difference (Final Values) = 19.18, 95% CI 2-sided [5.09 to 33.28]

13. Secondary Outcome: Proportion of Night Awakening Due to Asthma
Description: Change from baseline to Week 48 on proportion of night awakening due to asthma
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Mean (Standard Deviation); unit: Proportion of nights
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 210 | 193 | 195
Proportion of nights | -0.314 (0.366) | -0.380 (0.385) | -0.26 (0.344)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.964, Mixed Models Analysis; Model includes treatment, baseline proportion of nights with nocturnal awakenings, region, use of OCS, visit and visit by treatment; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.05 to 0.04]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis; [statistical method as in outcome 13, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.11 to -0.01]

14. Secondary Outcome: Mean Change From Baseline to Week 48 in ACQ-6 for Baseline Eosinophils >=300/uL
Description: ACQ-6 contains one bronchodilator question and 5 symptom questions. Questions are rated from 0 (totally controlled) to 6 (severely uncontrolled). Mean ACQ-6 score is the average of the responses. Mean scores of <=0.75 indicates well-controlled asthma, scores between 0.75 to <=1.5 indicate partly controlled asthma, and >1.5 indicates not well controlled asthma.
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 198 | 191 | 186
Scores on a scale | -1.33 (1.18) | -1.47 (1.05) | -1.12 (1.15)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.111, Mixed Models Analysis; Model includes treatment, baseline ACQ-6 score, region, use of OCS, visit and visit by treatment; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.34 to 0.04]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; Model includes treatment, baseline ACQ-6 score, region, use of OCS, visit and visit by treatment; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.48 to -0.10]

15. Secondary Outcome: Mean Change From Baseline to Week 48 in ACQ-6 for Baseline Eosinophils <300/uL
Description: as for outcome 14
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils <300/uL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 89 | 94 | 97
Scores on a scale | -0.77 (1.07) | -1.14 (1.11) | -0.89 (1.01)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.99, Mixed Models Analysis; Model includes treatment, baseline ACQ-6 score, region, use of OCS, visit and visit by treatment; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.27 to 0.27]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.107, Mixed Models Analysis; Model includes treatment, baseline ACQ-6 score, region, use of OCS, visit and visit by treatment; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.48 to 0.05]

16. Secondary Outcome: Pharmacokinetics of Benralizumab
Description: Mean PK concentrations at each visit
Time Frame: Baseline, week 4, week 4 day 6, week 8, week 16, week 24, week 32, week 40, week 48, week 56
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 399 | 391 | 0
ng/mL
  Baseline (n=395, 386) | NA (NA) — Value is less than lower limit of quantification | NA (NA) — Value is less than lower limit of quantification |
  Week 4 (n=393, 375) | 632.84 (152.14) | 629.89 (169.22) |
  Week 4 day 6 (n=54, 63) | 1368.98 (633.33) | 1273.7 (688.20) |
  Week 8 (n=377, 366) | 916.25 (142.53) | 881.57 (156.12) |
  Week 16 (n=358, 350) | 1024.26 (174.08) | 250.84 (228.25) |
  Week 24 (n=349, 344) | 926.62 (231.75) | 184.08 (298.92) |
  Week 32 (n=260, 267) | 853.67 (248.6) | 152.73 (394.18) |
  Week 40 (n=328, 333) | 967.15 (218.32) | 157.22 (364.6) |
  Week 48 (n=333, 333) | 864.37 (283.87) | 162.51 (352.46) |
  Week 56 (n=63, 67) | 51.7 (833.91) | 6.66 (321.88) |

17. Secondary Outcome: Immunogenicity of Benralizumab
Description: Anti-drug antibodies (ADA) responses at baseline and post baseline. Persistently positive is defined as positive at >=2 post baseline assessments (with >=16 weeks between the first and the last positive) or positive at last post baseline assessment. Transiently positive is defined as having at least one post baseline ADA positive assessment and not fulfilling the conditions of persistently positive.
Time Frame: Pre-treatment until end of follow-up
Population: Safety analysis set, note that 4 patients who were randomized to q.8 regimen treated with q.4 regimen. Thus 403 patients treated with q.4 rather than 399, 394 patients treated with q.8 rather than 398. However, data were only available for 402 patients in q.4, and 393 patients in q.8.
Measure: Number; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 402 | 393 | 407
Participants
  Positive at any visit (n=402, 393, 407) | 47 | 58 | 21
  Base- and post baseline positive (n=393, 381, 396) | 2 | 3 | 10
  Only post baseline positive (n=396, 389, 402) | 39 | 49 | 10
  Persistently positive (n=396, 389, 402) | 23 | 39 | 16
  Transiently positive (n=396, 389, 402) | 18 | 13 | 4
  Only baseline positive (n=399, 385, 401) | 6 | 6 | 1

18. Secondary Outcome: Extend of Exposure
Description: Extend of exposure is defined as duration of treatment in days
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Safety analysis set, note that 4 patients who were randomized to q.8 regimen treated with q.4 regimen. Thus 403 patients treated with q.4 rather than 399, 394 patients treated with q.8 rather than 398.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 403 | 394 | 407
Days | 285.86 (67.446) | 288.02 (66.683) | 289.38 (61.527)

19. Secondary Outcome: Mean Change From Baseline to Week 48 in AQLQ(S)+12
Description: AQLQ(S)+12 overall score is defined as the average of all 32 questions in the AQLQ(S)+12 questionnaire. AQLQ(S)+12 is a 7-point scale questionnaire, ranging from 7 (no impairment) to 1 (severe impairment). Total or domain score change of >=0.5 are considered clinically meaningful.
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 192 | 187 | 180
Scores on a scale | 1.44 (1.18) | 1.56 (1.17) | 1.25 (1.18)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.081, Mixed Models Analysis; Model includes covariates treatment, baseline AQLQ(S)+12 score, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.02 to 0.37]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Model includes covariates treatment, baseline AQLQ(S)+12 score, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [0.1 to 0.5]

20. Secondary Outcome: Mean Change From Baseline to Week 48 in EQ-5D-5L VAS
Description: EQ-5D-5L VAS is to rate current health status on a scale of 0-100, with 0 being the worst imaginable health state.
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 191 | 186 | 181
Scores on a scale | 13.5 (21.82) | 16.5 (23.66) | 12.5 (21.41)

21. Secondary Outcome: Mean Work Productivity Loss Due to Asthma
Description: WPAI+CIQ (Work Productivity and Activity Impairment plus Classroom Impairment Questionnaire) contains 10 questions. Work productivity loss is derived by sum of percentage of missed work due to asthma and product of percentage of actual working hours times degree of asthma affecting work productivity while working. Percentage of missed work due to asthma is calculated by number of hours missed work due to asthma divided by total number of hours missed work plus number of hours actually worked. The work productivity loss is only applicable to patients who employed, which is only subset of the study population.
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils >=300/uL for patients who employed
Measure: Mean (Standard Deviation); unit: Percent of productivity loss
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 85 | 79 | 76
Percent of productivity loss | 23.31 (24.169) | 26.11 (23.06) | 35.36 (24.537)

22. Secondary Outcome: Mean Productivity Loss Due to Asthma in Classroom
Description: WPAI+CIQ (Work Productivity and Activity Impairment plus Classroom Impairment Questionnaire) contains 10 questions. Classroom productivity loss is derived by sum of percentage of missed classes due to asthma and product of percentage of actual hours attending classes times degree of asthma affecting classroom productivity. Percentage of missed classes due to asthma is calculated by number of hours missed classes due to asthma divided by total number of hours missed classes plus number of hours actually attending classes. This is only applicable to patients who attending classes
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils >=300/uL who attending classes
Measure: Mean (Standard Deviation); unit: Percent of productivity loss
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 8 | 6 | 18
Percent of productivity loss | 30.97 (25.311) | 27.17 (38.456) | 49.1 (25.801)

23. Secondary Outcome: Number of Participants That Utilized Health Care Resources
Time Frame: Immediately following the first administration of study drug through Study Week 48.
Population: Full analysis set, Baseline eosinophils >=300=/uL
Measure: Number; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 275 | 267 | 267
Participants
  Hospitalizations | 14 | 12 | 20
  Emergency department visits | 20 | 10 | 26
  Unscheduled outpatient visits | 77 | 87 | 109
  Home visits | 2 | 1 | 3
  Telephone calls | 46 | 41 | 62
  Ambulance transports | 6 | 3 | 9

24. Secondary Outcome: Patient and Clinician's Responder Assessment to Treatment
Description: CGIC (Clinical global impression of change), and PGIC (Patient global impression of change) are overall evaluation of response to treatment, conducted separately by investigator and patient using 7-point rating scale, ranging from 1 (very much improved), to 7 (very much worse). This is additional measures collected after second Amendment, thus not all patients had data to be analyzed.
Time Frame: Immediately following the first administration of study drug through Study Week 48
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Number; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 275 | 267 | 267
Participants
  CGIC improved | 80 | 76 | 88
  CGIC much improved | 59 | 58 | 58
  CGIC very much improved | 18 | 12 | 5
  CGIC total responder | 157 | 146 | 151
  PGIC improved | 84 | 80 | 91
  PGIC much improved | 55 | 58 | 65
  PGIC very much improved | 26 | 19 | 11
  PGIC total responder | 165 | 157 | 167

ADVERSE EVENTS:
Description: There were 400 patients randomized to Benra q.4, and 398 patients randomized to Benra q.8. One patient in Benra q.4 was never treated. In addition, 4 patients who were randomized to q.8 group, but were treated with q.4 schedule. So 403 patients were treated with q.4 regimen, and 394 patients were treated with q.8 regimen.
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Serious Adverse Events (participants affected / at risk) | 51/403 | 54/394 | 58/407
Other Adverse Events (participants affected / at risk) | 214/403 | 199/394 | 219/407
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab 30 mg q.4 Weeks (N=403) | Benralizumab 30 mg q.8 Weeks (N=394) | Placebo (N=407)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1)
Allergic granulomatous angiitis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bullous impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (3) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Adenolymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Aphonia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral venous thrombosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 23 (29) | 24 (33) | 32 (42)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab 30 mg q.4 Weeks (N=403) | Benralizumab 30 mg q.8 Weeks (N=394) | Placebo (N=407)
Nausea (Gastrointestinal disorders) | 8 (12) | 12 (14) | 8 (9)
Pyrexia (General disorders) | 16 (21) | 12 (19) | 8 (8)
Acute sinusitis (Infections and infestations) | 10 (11) | 13 (14) | 11 (15)
Bronchitis (Infections and infestations) | 27 (28) | 19 (22) | 30 (41)
Gastroenteritis (Infections and infestations) | 10 (16) | 12 (14) | 6 (6)
Influenza (Infections and infestations) | 15 (19) | 19 (21) | 23 (31)
Nasopharyngitis (Infections and infestations) | 47 (62) | 47 (69) | 49 (64)
Pharyngitis (Infections and infestations) | 17 (21) | 23 (24) | 14 (20)
Rhinitis (Infections and infestations) | 16 (17) | 10 (11) | 15 (17)
Sinusitis (Infections and infestations) | 18 (23) | 22 (34) | 29 (43)
Upper respiratory tract infection (Infections and infestations) | 45 (74) | 32 (51) | 37 (73)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (13) | 18 (20) | 12 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 8 (9) | 15 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 13 (13) | 5 (6)
Headache (Nervous system disorders) | 31 (38) | 37 (61) | 21 (28)
Asthma (Respiratory, thoracic and mediastinal disorders) | 48 (64) | 27 (38) | 60 (102)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 13 (14) | 11 (15)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 12 (12) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.